CLINICAL TRIAL: NCT00412919
Title: A Prospective, Single-Arm, 2-Stage, Open-label, Phase II Trial of Azacitidine in Relapsed and Refractory Multiple Myeloma.
Brief Title: Study of Azacitidine to Treat Relapsed or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AH213/06
Record Dates: First submitted 2006-12-17; First posted 2006-12-19 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2006-12

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Relapsed; Refractory
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Recurrence | interventions — Azacitidine

INTERVENTIONS:
Drug: Azacitidine

SUMMARY:
This is a Phase II trial evaluating the overall response rate, safety and tolerability to azacitidine in patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is an incurable disease with an annual incidence of 14,000 new cases in the US alone. Despite initial sensitivity to corticosteroids, chemotherapy and radiotherapy, relapse is inevitable and there is a median survival of only 2.5 to 3 years. The use of autologous stem cell transplantation (SCT) has improved the duration of disease remission for younger patients but still only results in a median survival of 5 - 6 years.

Since the early 1970s, azacitidine has been investigated for the treatment of acute leukemia. More recently it has been investigated in the treatment of patients with myelodysplastic syndrome (a pre-leukaemic condition). It has been shown to prolong the time to development of acute myeloid leukaemia (AML) or death and has now been approved for use in these patients.

Azacitidine is a cytotoxic drug and is directly toxic to cells, preventing their reproduction or growth. It is also able to cause cells to undergo the process whereby they mature into normal cells. The Myeloma Research Group at The Alfred Hospital has looked at the effect of azacitidine on human myeloma cell lines in the laboratory. Azacitidine was found to prevent both cell growth and causes cell death. In mouse models with multiple myeloma azacitidine prolonged their survival.

The primary aim of this study is to determine the effectiveness of azacitidine in treating patients with multiple myeloma. The other aims of this study are to see whether treating patients with azacitidine extends the time that their myeloma is under control, to determine the number of cycles of azacitidine required to first achieve a response and to determine how safe and tolerable azacitidine is in treating multiple myeloma.

In the first stage a total of 14 people will participate in this project. If in this group of patients azacitidine is shown to be effective as a treatment against multiple myeloma then a further 10 patients will be invited to participate.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of MM as per IMWG criteria
* age greater than 17 years
* have received at least 2 but no more than 4 prior lines of therapy
* have failed to respond to the most recently administered anti-MM therapy or have demonstrably progressive disease as defined by accepted standard criteria
* have a life expectancy of at least 3 months
* ECOG performance status < 3
* at registration haematological values within the following limits:

  1. absolute neutrophil count (ANC) > 1.0 x 109/L
  2. platelet count > 50 x 109/L unsupported
* At registration biochemical values within the following limits

  1. Bilirubin < 1.5 x upper limit of normal (ULN) and transaminases < 2 x ULN unless considered secondary to hepatic myelomatous infiltration
  2. Serum creatinine < 0.19mMol/L
* Written informed consent
* Must agree to use adequate contraceptive measures if indicated. Specifically, women of childbearing potential (WOCBP) may participate provided they meet the following conditions:

  1. Agree to use at least 2 effective contraceptive methods throughout the study and for 30 days following the study
  2. Have a negative serum pregnancy test within 24 hours of commencing on study medication
  3. Male participants with female partners that are WOCBP must agree to use 2 effective contraceptive methods throughout the study and for 30 days following the study

Exclusion Criteria:

* Patients with monoclonal gammopathy of undetermined significance (MGUS) or indolent/smouldering MM
* Known or suspected hypersensitivity to AZA or mannitol
* Patients whose general condition makes them unsuitable for intensive treatment e.g. significant cardiac or pulmonary disease
* Active infections or other illnesses that precludes chemotherapy administration or patient compliance
* Active viral infection with known human immunodeficiency virus (HIV) or viral hepatitis type B or C
* Pregnant or lactating women

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-12; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Overall response rate

SECONDARY OUTCOMES:
time to progression
duration of response
number of cycles of azacitidine required to first achieve a response
progression free survival
safety
tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Spencer, Assoc. Prof, Study Chair
Locations (1):
- The Alfred Hospital, Melbourne, Victoria, Australia